CLINICAL TRIAL: NCT07316075
Title: Multicenter Study on Cardiovascular and Metabolic Complications in Patients With Biochemically Silent Pheochromocytomas and Paragangliomas
Status: Enrolling by invitation | Type: Observational
Sponsor: Laikο General Hospital, Athens (Other)
Responsible Party: Principal Investigator, Anna Angelousi, Associate Professor, Laikο General Hospital, Athens
Other Study IDs: 2240/12.02.2025
Record Dates: First submitted 2025-12-07; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Abnormalities; Arterial Blood Pressure; Heart Rate; Congestive Heart Failure Chronic; Coronary Syndrome; Cerebrovascular Disease; Myocarditis, Pericarditis; Hyperlipidaemia; Diabete Mellitus
Keywords: pheochromocytoma; paraganglioma; cardiovascular risk; cerebrovascular risk; blood pressure; coronary syndrome; heart rate; metabiolic syndrome; hypelipidemia; diabetes
MeSH Terms: conditions — Cardiovascular Abnormalities; Angina, Unstable; Cerebrovascular Disorders; Myocarditis; Pericarditis; Hyperlipidemias; Diabetes Mellitus; Pheochromocytoma; Paraganglioma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with biochemically silent PPGLs: Patients with non-detectable levels of metanephrines/normetanephrines in the blood or in the urine via LC-MS.
- Controls ( healthy individuals): Healthy individuals with normal adrenal gland
- Patients with secreting PPGLs: Patients with measurable levels of metanephrines or normetanephrines in the blood or urine ( > 2-fold) via LC-MS

SUMMARY:
The aim of the study is to characterise the cardiovascular and metabolic complications pre- and post-surgery of patients with biochemically negative PPGL and to compare them with normal individuals and patients with secreting PPGLs age and sex matched.

DETAILED DESCRIPTION:
Pheochromocytomas (PHEO) and Paragangliomas (PGL) represent a group of tumors associated with increased cardiometabolic morbidities and mortality. The secretory components of PHEOs/PGLs are well-established risk factors for cardiovascular events and the Endocrine Society Clinical Practice Guidelines have implemented specific instructions for their management and their follow-up. However, data regarding the cardiovascular risk in PHEOs and PGLs asymptomatic patients with the normal biochemical profile are sparse and debating. The incidence of cardiovascular complications and the long-term morbidity in this group of patients is not well-characterized complicating the therapeutic approach or the necessity of pre-operative a-blockade as well as the optimal follow-up, regarding the duration and the need for cardiovascular examination.

Aim Primary outcome v To characterize the cardiovascular and metabolic complications of patients with biochemically negative PPGLs and to compare them with individuals age and sex-matched with normal adrenals (controls) as well as with patients with secreting PHEOs/PGLs.

Secondary outcome v To study also the sub-mentioned parameters post-treatment

ELIGIBILITY:
Inclusion Criteria:

* All PHEOs/PGLs patients should be asymptomatic, with confirmed histopathological analysis for those who had surgery or with positive specific imaging functional studies (MIBG, 68Ga DOTATATE, Octreoscan, Tektrotyde)
* Data about the plasma or urine levels of catecholamines, normetanephrines, metanephrines and methoxytyramine (for PGL) levels should be available for every patient and should be lower than the upper normal values measured with LC-MS (supplementary data about CgA, NSE levels can be also included)
* Available data for the "required" cardiovascular paraclinical or metabolic parameters should be available pre-surgery or at the time of diagnosis or at follow-up for the "not operable" tumors as well as post any treatment

Exclusion Criteria:

* Patients with ambiguous diagnosis of PHEOs/PGLs (absence of histological report and non-specific imaging findings)
* Catecholamines, normetanephrines and metanephrines (and methoxytyramine levels for PGL) levels higher than the upper limit range
* No available data of the required parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any adult patient with a confirmed histopathological or imaging diagnosis of PPGL (biochemical silent vs secreting)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2027-02-25 (Estimated)

PRIMARY OUTCOMES:
Changes in arterial blood pressure (BP) in mmHg before and after any therapeutic intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  Mean Systolic and diastolic BP (x3) in mmHg before and after any therapeutic intervention or follow-up
Changes in the heart rate (pulsation/min) before and after any therapeutic intervention or follow-up | Baseline at diagnosis and 6 months post any intervention or follow-up
  Mean heart rate before and after any therapeutic intervention or follow-up
Changes in the fraction of ejection of the heart estimated by cardiac triplex before and after any treatment | Baseline at diagnosis and 6 months post any intervention or follow-up
  Echocardiogram and estimation of fraction of ejection before and after any treatment or follow-up
Incidence (number) and characterisation of coronary syndrome (angina, cardiac infarction) before and after any intervention or follow-up | Baseline at diagnosis and 6 months post any intervention or follow-up
  Incidence of an episode of coronary syndrome, like angina or cardiac infarction and evaluation of the electrocardiogram (changes of ST waves or Q waves or Left blovk branch) and signs of ventricule hypokinesia or akinesia in the heart triplex before and after any treatment or follow-up
Incidence of cerebrovascular event permanent or transient | Baseline at diagnosis and 6 months post any intervention or follow-up
  Incidence of cerebrovascular disease, permanent or transient, and evaluation with cerebral MRI before and after any therapeutic intervention
Incidence of myocarditis before and after any therapeutic intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  episode of myocarditis based on increased troponine, cardiac MRI and heart triplex before and after any intervention

SECONDARY OUTCOMES:
Changes in the levels of blood Hb1Ac before and after any therapeutic intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  Measurement of Hb1AC % in the blood
Changes in the concentrations of cholesterol, LDL and HDL in the blood before and after any intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  Measurement of blood cholesterol in mg/dl, HDL in mg/dl and LDL in mg/dl before and after any therapeutic intervention

OTHER OUTCOMES:
Changes of the Intima-Media Thickness and of Atheromatous Plaque before and after any intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  Triplex of carotides with measurement in mm of Intima-Media Thickness and of Atheromatous Plaque (appearance, surface)before and after any intervention
Changes of proBNP levels in the blood before and after any intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  Mesurement of proBNP at blood analysis (pg/ml)
Changes in troponine levels in the blood before and after any therapeutic intervention | Baseline at diagnosis and 6 months post any intervention or follow-up
  Measurement of troponine levels (ng/ml) in the blood

CONTACTS AND LOCATIONS:
Locations (1):
- NKUA, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided
Personal protection data

REFERENCES:
- [Background] Zhou J, Xuan H, Miao Y, Hu J, Dai Y. Acute cardiac complications and subclinical myocardial injuries associated with pheochromocytoma and paraganglioma. BMC Cardiovasc Disord. 2021 Apr 21;21(1):203. doi: 10.1186/s12872-021-02013-6. PMID 33882857
- [Background] Kumar A, Pappachan JM, Fernandez CJ. Catecholamine-induced cardiomyopathy: an endocrinologist's perspective. Rev Cardiovasc Med. 2021 Dec 22;22(4):1215-1228. doi: 10.31083/j.rcm2204130. PMID 34957765
- [Background] Szatko A, Glinicki P, Gietka-Czernel M. Pheochromocytoma/paraganglioma-associated cardiomyopathy. Front Endocrinol (Lausanne). 2023 Jul 13;14:1204851. doi: 10.3389/fendo.2023.1204851. eCollection 2023. PMID 37522121
- [Background] Y-Hassan S, Falhammar H. Cardiovascular Manifestations and Complications of Pheochromocytomas and Paragangliomas. J Clin Med. 2020 Jul 30;9(8):2435. doi: 10.3390/jcm9082435. PMID 32751501
- [Background] Constantinescu G, Preda C, Constantinescu V, Siepmann T, Bornstein SR, Lenders JWM, Eisenhofer G, Pamporaki C. Silent pheochromocytoma and paraganglioma: Systematic review and proposed definitions for standardized terminology. Front Endocrinol (Lausanne). 2022 Oct 17;13:1021420. doi: 10.3389/fendo.2022.1021420. eCollection 2022. PMID 36325453